CLINICAL TRIAL: NCT07249905
Title: A Phase 1/2 Clinical Study Evaluating MDX2003 in Participants With Relapsed, Progressive, or Refractory B-Cell Malignancies
Brief Title: This Study is Designed to Characterize the Safety, Tolerability, and Anti-tumor Activity of MDX2003 in Patients With Different Types of Lymphoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModeX Therapeutics, An OPKO Health Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDX-2003-101
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Lymphoma; Waldenström Macroglobulinemia (WM); DLBCL - Diffuse Large B Cell Lymphoma; PMBCL; HGBCL; FL Lymphoma; Lymphoplasmacytic Lymphoma; Follicular Lymphoma (FL)
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation- Part A (Experimental): Participants with B-cell malignancies will receive MDX2003 as an intravenous (IV) infusion.
  Interventions: Drug: MDX2003
- Indication Optimization- Part B (Experimental): Participants with select B-cell malignancies will receive MDX2003 as an intravenous (IV) infusion.
  Interventions: Drug: MDX2003

INTERVENTIONS:
Drug: MDX2003 — MDX2003 intravenous infusion

SUMMARY:
This study is designed to characterize the safety, tolerability, and anti-tumor activity of MDX2003 in patients with different types of lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age.
* Participant has a confirmed diagnosis of large B-cell lymphoma (including DLBCL, high-grade B-cell lymphoma [HGBCL], primary mediastinal B-cell lymphoma [PMBCL], etc), FL, MCL, marginal zone lymphoma, transformation of indolent B-cell lymphoma, or lymphoplasmacytic lymphoma, including Waldenstrom macroglobulinemia.
* Participant has relapsed or progressed on at least 2 prior lines of therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* All participants must have measurable disease via computed tomography (CT), magnetic resonance imaging (MRI), or positron emission tomography (PET)-CT.
* Documented CD19 or CD20 positivity of their B-cell neoplasm based on any representative pathology report from the past 3 months.
* Adequate hematologic, hepatic and renal function.
* All contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH).
* Unresolved toxicities from previous anticancer therapy.
* Primary central nervous system (CNS) lymphoma or known CNS involvement with lymphoma.
* Active medical condition requiring chronic systemic steroid use (>10 mg/day prednisone or equivalent of >140 mg over the last 14 days) or immunosuppressive therapy, within 6 months prior to the first dose of MDX2003.
* Known positivity with human immunodeficiency virus (HIV), known active hepatitis B or C, or uncontrolled chronic or ongoing infection requiring intravenous treatment.
* Participant has a history of allogenic tissue or solid organ transplant, with the exception of corneal transplants.
* Known hypersensitivity to allopurinol or rasburicase.
* Participant has a seizure disorder requiring therapy at the time of screening (such as steroids or anti-epileptics).
* Participant is not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Part A only- Identify the Maximum Tolerated Dose (MTD) for expansion for further development of MDX2003 | 28 days
  Maximum Tolerated Dose is determined following the evaluation of MDX2003 safety, including the incidences of dose-limiting toxicities (DLTs), MDX2003 anti-tumor activity, and MDX2003 pharmacokinetics/pharmacodynamics.
All Study Parts: Adverse Events (AEs) | Baseline until 90 days after the participant has the last dose of MDX2003
  Incidence and severity of adverse events (AEs) and serious AEs (SAEs), including changes in clinical laboratory parameters, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0 or American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading criteria, including changes in clinical laboratory parameters.
Part B only- Assess the preliminary anti-lymphoma activity of MDX2003 | From date of enrollment until the end of treatment, up to approximately 6 months
  Objective response rate is defined as the proportion of patients who achieve a complete response (CR) or partial response (PR) per Lugano Classification.

SECONDARY OUTCOMES:
All Study Parts: Measure of terminal half-life (t1/2) of MDX2003 | 6 months
  Characterize pharmacokinetic (PK) parameter t1/2 after intravenous infusion of MDX2003.
All Study Parts: Measure of area under the serum concentration-time curve (AUC) of MDX2003 | 6 months
  Characterize pharmacokinetic (PK) parameter AUC after intravenous infusion of MDX2003.
All Study Parts: Measure of time to maximum concentration (Tmax) of MDX2003 | 6 months
  Characterize pharmacokinetic (PK) parameter Tmax after intravenous infusion of MDX2003.
All Study Parts: Measure of maximum serum concentration (Cmax) of MDX2003 | 6 months
  Characterize pharmacokinetic (PK) parameter Cmax after intravenous infusion of MDX2003.
All Study Parts: Measure of volume of distribution (Vd) of MDX2003 | 6 months
  Characterize pharmacokinetic (PK) parameter Vd after intravenous infusion of MDX2003.
All Study Parts: Measure of system clearance of MDX2003 | 6 months
  Characterize pharmacokinetic (PK) parameter of system clearance after intravenous infusion of MDX2003.
All Study Parts: Evaluation of MDX2003 immunogenicity | 6 months
  The presence and persistence of anti-MDX2003 antibodies.

IPD SHARING:
Plan to Share IPD: No